CLINICAL TRIAL: NCT00691444
Title: Melatonin Studies of Blind Children
Brief Title: Blind Child Melatonin Treatment Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unique provision in the American Recovery and Reinvestment Act prevented approval of second year no-cost-extension in which completion of analyses were planned.
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eIRB 1251; R01HD042125 (NIH)
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Blindness
Keywords: melatonin; circadian rhythms; sleep
MeSH Terms: conditions — Blindness | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Subjects will be given up to 0.5 mg daily. If the treatment works, the dose will be reduced gradually until the lowest, effective dose is identified. If the treatment is unsuccessful, the subject will be taken off treatment and later enrolled in a different treatment plan.
  Interventions: Dietary Supplement: Melatonin
- 2 (Experimental): Subjects will be given up to 10 mg daily. If the treatment works, the dose will be reduced gradually until the lowest, effective dose is identified. If the treatment is unsuccessful, the subject will be taken off treatment and later enrolled in a different treatment plan.
  Interventions: Dietary Supplement: Melatonin
- 3 (Experimental): Subjects will be given up to 20 mg daily. If the treatment works, the dose will be reduced gradually until the lowest, effective dose is identified. If the treatment is unsuccessful, the subject will be taken off treatment and later enrolled in a different treatment plan.
  Interventions: Biological: Melatonin

INTERVENTIONS:
Dietary Supplement: Melatonin — Subjects will be given up to 0.5 mg daily.
  0.005-20 mg, daily, up to 5 years (the exact duration depends on each subjects response to the dose and the specifics of their circadian rhythm patterns).
  Arms: 1
Dietary Supplement: Melatonin — Subjects will be given up to 10 mg daily.
  0.005-20 mg, daily, up to 5 years (the exact duration depends on each subjects response to the dose and the specifics of their circadian rhythm patterns).
  Arms: 2
Biological: Melatonin — Subjects will be given up to 20 mg daily.
  0.005-20 mg, daily, up to 5 years (the exact duration depends on each subjects response to the dose and the specifics of their circadian rhythm patterns).
  Arms: 3

SUMMARY:
The primary focus of this five-year study will be to optimize the melatonin dosing regimen for synchronizing the body clocks of blind children to the 24-hour day.

DETAILED DESCRIPTION:
We intend to study as many as 26 blind children through up to three melatonin treatment regimens, all of which involve a dose step-down in which the melatonin dose will be reduced gradually to find the lowest effective dose. The 3 treatment plans differ only in the start dose. Successfully treated subjects (of one treatment plan) will enter a one-year intensive assessment of the safety and efficacy of melatonin treatment in which the subject will take the same dose for one year and complete biweekly assessments of efficacy and side-effects. The final phase of the study involves a placebo discontinuation, in which the subject's circadian rhythm will be returned to the baseline rhythm (this may take up to 6 months for some subjects).

ELIGIBILITY:
Inclusion Criteria:

* Children and adults 5 to 20 years old
* Blindness for at least one year, verified by an ophthalmologic exam
* Ability to comply with the requirements of the experimental protocol
* And no clinically significant abnormalities (other than blindness) on a general physical examination.
* Subjects must be competent to sign informed consent if age 18 or older. Parents and subjects will be interviewed together and, when appropriate (for example, subject is age 18 or older), separately as well.

Exclusion Criteria:

* Abnormal heart, liver or kidney function; intractable seizure disorders
* Significant laboratory abnormalities on CBC, Comprehensive Metabolic set, or UA (dip stick method)
* Pregnancy; sexual activity in post-pubertal females not using a recognized and valid contraceptive method
* A current Axis I psychiatric or substance abuse disorder according to the DSM-IV Manual ; OR
* External demands that limit the ability to maintain a regular schedule, e.g. night shift work.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2002-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred J Lewy, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Sleep and Mood Disorders Lab, Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Lewy AJ, Emens J, Jackman A, Yuhas K. Circadian uses of melatonin in humans. Chronobiol Int. 2006;23(1-2):403-12. doi: 10.1080/07420520500545862. PMID 16687313
- [Background] Stores G, Ramchandani P. Sleep disorders in visually impaired children. Dev Med Child Neurol. 1999 May;41(5):348-52. doi: 10.1017/s0012162299000766. No abstract available. PMID 10378763

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- 0.5mg Melatonin: Subjects will be given up to 0.5 mg daily. If the treatment works, the dose will be reduced gradually until the lowest, effective dose is identified. If the treatment is unsuccessful, the subject will be taken off treatment and later enrolled in a different treatment plan.
  Melatonin: Subjects will be given up to 0.5 mg daily.
  0.005-20 mg, daily, up to 5 years (the exact duration depends on each subjects response to the dose and the specifics of their circadian rhythm patterns).
- 10mg Melatonin: Subjects will be given up to 10 mg daily. If the treatment works, the dose will be reduced gradually until the lowest, effective dose is identified. If the treatment is unsuccessful, the subject will be taken off treatment and later enrolled in a different treatment plan.
  Melatonin: Subjects will be given up to 10 mg daily.
  0.005-20 mg, daily, up to 5 years (the exact duration depends on each subjects response to the dose and the specifics of their circadian rhythm patterns).
- 20mg Melatonin: Subjects will be given up to 20 mg daily. If the treatment works, the dose will be reduced gradually until the lowest, effective dose is identified. If the treatment is unsuccessful, the subject will be taken off treatment and later enrolled in a different treatment plan.
  Melatonin: Subjects will be given up to 20 mg daily.
  0.005-20 mg, daily, up to 5 years (the exact duration depends on each subjects response to the dose and the specifics of their circadian rhythm patterns).
Period: Overall Study
Arm/Group | 0.5mg Melatonin | 10mg Melatonin | 20mg Melatonin
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5mg Melatonin | 10mg Melatonin | 20mg Melatonin | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Circadian Phase Marker, as Measured by the Melatonin Levels in Serial Salivary and/or Plasma Samples.
Time Frame: biweekly throughout the entire study
Population: as for baseline characteristics
Arm/Group | 0.5mg Melatonin | 10mg Melatonin | 20mg Melatonin
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Durability and Toxicity Side Effects Questionnaire
Time Frame: 1 year
Population: as for baseline characteristics
Arm/Group | 0.5mg Melatonin | 10mg Melatonin | 20mg Melatonin
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | 0.5mg Melatonin | 10mg Melatonin | 20mg Melatonin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Analyses were not completed because, a unique provision in the American Recovery and Reinvestment Act (ARRA) of 2009 funding source unexpectedly prevented approval of a second year no-cost-extension in which completion of analyses were planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No